CLINICAL TRIAL: NCT00121888
Title: Randomized Trial of Paroxetine-CR for the Treatment of Patients With Post Traumatic Stress Disorder Remaining Symptomatic After Initial Exposure Therapy
Brief Title: Trial of Paroxetine-CR for the Treatment of Patients With Post Traumatic Stress Disorder Remaining Symptomatic After Initial Exposure Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Naomi M. Simon, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002-P-001879
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: post traumatic stress disorder; Prolonged Exposure Therapy; pharmacotherapy; double-blind; Anxiety Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy
Drug: Paroxetine-CR

SUMMARY:
The purpose of the study is to evaluate the effectiveness and tolerability of controlled-release paroxetine (Paxil-CR) compared to placebo (an inactive substance) for individuals who continue to have symptoms of post traumatic stress disorder (PTSD) despite receiving prolonged exposure therapy.

DETAILED DESCRIPTION:
Post Traumatic Stress Disorder (PTSD) is common in the general population with the National Comorbidity Survey reporting a lifetime prevalence of about 8% in the United States (Kessler, et al 1995). PTSD is associated with marked symptomatic distress as well as significant impairment, dysfunction and reduction in overall quality of life (Kessler, 2000). Both pharmacotherapeutic interventions, including serotonin selective reuptake inhibitors (SSRIs), and psychosocial interventions such as cognitive-behavior therapy (CBT) have demonstrated efficacy for PTSD (Davidson, 2001; Foa, 2000) However, although these interventions can be helpful, many patients remain symptomatic despite initial treatment. There is little data available to guide practice regarding the efficacy of "next step" strategies for patients remaining symptomatic despite treatment.

In this study the researchers will examine the relative efficacy of the addition of the SSRI, paroxetine-CR, compared to placebo for patients remaining symptomatic despite a brief and intensive course of CBT.

This is a two phase, 14-16 week research study in which participants who remain symptomatic at the end of one phase (4-6 weeks) enter into the next phase. In phase I, all participants receive prolonged exposure (PE) therapy. Participants who continue to have significant distress because of posttraumatic stress disorder after 8 sessions of therapy will enter Phase II. In Phase II subjects will receive 5 more sessions of PE therapy and be randomly assigned (by chance, like a flip of a coin) to receive paroxetine-cr (Paxil-CR) or placebo (contains no active medication). Participants receive this combined treatment over the next 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age with a primary (the condition that is most central to the patient's current distress) psychiatric diagnosis of PTSD as defined by DSM-IV criteria.
* Patients must have remained symptomatic (CGI-S > 3) and a score of at least 6 on the Short PTSD Rating Interview (SPRINT) after a minimum of 7 sessions of PE (delivered within 6 weeks) to be eligible for randomized treatment.

Exclusion Criteria:

* Patients will be excluded from the study for serious medical illness or instability for which hospitalization may be likely within the next three months.
* Pregnant or lactating women or those of childbearing potential not using medically accepted forms of contraception will be excluded.
* Concurrent use of other psychotropic medications; all psychotropic medications (excluding benzodiazepines) must be stopped at least one week prior to entry into the initial PE phase of the study. Patients may remain on concomitant benzodiazepines (<2 mg/d clonazepam or its equivalent), as long as the benzodiazepine therapy was initiated at least 2 months prior to randomization and at a constant dose for >4 weeks prior to randomization; the dose will be held constant through the study.
* Lifetime diagnosis of schizophrenia or any other psychosis, mental retardation, organic mental disorders, or bipolar disorder; obsessive-compulsive disorder, eating disorders, cutting or other significant self-injurious behavior or alcohol/substance abuse disorders within the last 6 months, are study exclusions. Patients with a current primary diagnosis of major depression, dysthymia, social anxiety disorder and generalized anxiety disorder are excluded - the presence of these disorders is permissible as long as the PTSD is the predominant disorder.
* Patients with a history of hypersensitivity or poor response to paroxetine are excluded. Concurrent dynamic or supportive psychotherapy is permitted as long as it is has been ongoing for at least 2 months prior to onset of study entry.
* Patients with current compensation or legal actions related to the effects of the trauma, or those with an ongoing relationship with their assailant.
* Patients with a positive toxicology screen at baseline consistent with evidence of current substance abuse or dependence as determined by clinical interview.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of post traumatic stress disorder

SECONDARY OUTCOMES:
Clinical global improvement

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Simon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: The Center for Anxiety and Traumatic Stress Disorders at Massachusetts General Hospital — http://www.mghanxiety.org